CLINICAL TRIAL: NCT04689256
Title: Pilot Randomized Controlled Study of the Impact of MedRhythms' MR-010 in Acute Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to lower than expected recruitment
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: MedRhythms, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H00021940
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Stroke, Acute
Keywords: rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- MR-010 walking therapy (Experimental): Subjects will use the MR-010 three times a week for 30 minutes per session for 90 days. Subjects will undergo a 10-meter walk test bi-weekly and at 45 and 90 days.
  Interventions: Device: MR-010
- Standard of Care (No Intervention): Subjects will undergo a 10-meter walk test bi-weekly for 90 days and at 45 and 90 days

INTERVENTIONS:
Device: MR-010 — MR-010 includes a patient application and sensors with commercially available headphones and smartphones. Sensors are placed on the subject's shoes and measure gait metrics. The algorithm uses data from the sensors to inform changes made to the audio cues. These cues, which are embedded in time-shifted music, are delivered back to the users who aim to walk to the beat.
  Arms: MR-010 walking therapy

SUMMARY:
The purpose of this clinical pilot study is to evaluate the effects of the MR-010 on tolerability, biomechanics and walking speed in the acute stroke care setting in addition to its impact on length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older.
* Must be able to read and speak English fluently.
* Be within 24 hours from admission for confirmed stroke event.
* Currently able to walk at a speed greater or equal to 0.4m/s, but less than 1.0m/s, as determined by a 10-meter walk test for comfortable walking speed (the average of three trials).
* Demonstrates some level of asymmetry in gait.
* Is expected to be discharged from the acute care setting requiring physical therapy per standard of care and participant has verbally committed to receiving at least one therapy session.
* Able and willing to consent with proposed study schema (verbal commitment), including consent to participate in communication with the treating clinician (as needed) during the study period.
* Score ≤1 on question 1b and a 0 on question 1c on the NIH Stroke Scale.
* Able to safely participate in protocol-defined walking therapy sessions of 30-minute duration as determined by the Investigator.

Exclusion Criteria:

* Participant unable or unwilling to provide informed consent.
* Has a known history of neurologic (excluding stroke) injury.
* Has severe aphasia and/or a speech/language disorder, limiting ability to express needs and comprehend instructions.
* Has an external lower limb prosthetic ("artificial limb").
* Has a hearing impairment.
* Had orthopedic surgery in the last year.
* Has co-morbidities that prevent participation in exercise (for example: musculoskeletal, cardiovascular, pulmonary and neurological - other than stroke).
* Vulnerable populations as deemed inappropriate for study by site Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Silver, MD, Principal Investigator — UMass Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited in hospital after confirmed diagnosis of acute stroke from 11/03/2021 to 11/27/2022. Study terminated due to lower than expected recruitment
Pre-assignment Details: Patients included following diagnosis of acute stroke
Period: Overall Study
Arm/Group | MR-010 Walking Therapy | Standard of Care
Started | 2 | 2
Completed | 0 | 2
Not Completed | 2 | 0
Not completed — Participants declined to participate in the interventions per protocol | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MR-010 Walking Therapy | Standard of Care | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 66.5 [66 to 67] | 67.5 [65 to 70] | 67 [65 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Gait Speed (m/s)
Description: Change in gait speed (m/s) from baseline to study completion as measured by a 6 meter walking test.
Time Frame: 90 days
Population: No subjects completed the at home 6 Meter Walking Test. Therefore, no data was collected for this outcome measure.
Arm/Group | MR-010 Walking Therapy | Standard of Care
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Adherence to MR-010 Therapy Schedule
Description: Adherence to the MR-010 therapy schedule is measured by the number of participants who completed scheduled sessions (3 times per week for 12 weeks)
Time Frame: 90 days
Population: Data for this outcome was only intended to be collected and measured for participants in the MR-010 walking therapy group. As no participants completed the MR-101 walking therapy intervention, no data was collected.
Arm/Group | MR-010 Walking Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Length of Stay
Description: Median length of stay in acute stroke hospital
Time Frame: Duration of hospital stay, up to 14 days
Measure: Median (Full Range); unit: days
Arm/Group | MR-010 Walking Therapy | Standard of Care
Number analyzed (Participants) | 2 | 2
days | 3 [2 to 4] | 3 [2 to 4]

4. Secondary Outcome: Readmission to Hospital
Description: Percent of readmission to hospital following discharge
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | MR-010 Walking Therapy | Standard of Care
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | MR-010 Walking Therapy | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
In this study, the intervention group opted not to use the devices or participate in interventions or self-measured data as outlined in the protocol. Further, the study was closed early due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-07-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT04689256/Prot_001.pdf